CLINICAL TRIAL: NCT02323737
Title: Cisplatin Combined With Irinotecan or Etoposide for Untreated Extensive-stage Small Cell Lung Cancer: a Multicenter Randomized Control Clinical Trial
Brief Title: Phase II Study of Irinotecan and Cisplatin in Extensive-stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-022
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irinotecan and cisplatin (Active Comparator): The IP regimen consisted of at most 6 cycles of irinotecan 65 mg/m2 of body-surface area on days 1, 8 and cisplatin 75mg/m2 of body-surface area on day 1.
  Interventions: Drug: Irinotecan and cisplatin
- Etoposide and Cisplatin (Active Comparator): The EP regimen consisted of at most 6 cycles of etoposide 100 mg/m2 of body-surface area from day 1 to 3 and cisplatin 75mg/m2 of body-surface area on day 1.
  Interventions: Drug: Etoposide and cisplatin

INTERVENTIONS:
Drug: Irinotecan and cisplatin
  Arms: Irinotecan and cisplatin
Drug: Etoposide and cisplatin
  Arms: Etoposide and Cisplatin

SUMMARY:
Patients with untreated extensive-stage small cell lung cancer(SCLC) were randomly assigned to receive either irinotecan/cisplatin (IP) or etoposide/cisplatin(EP), The association of efficacy and toxicity of IP regimen was analyzed.

DETAILED DESCRIPTION:
This is a randomized, multicenter study. Patients are randomized to irinotecan/cisplatin (IP) or etoposide/cisplatin (EP) treatment arms. The IP regimen consisted of at most 6 cycles of irinotecan 65 mg/m2 of body-surface area on days 1, 8 and cisplatin 75mg/m2 of body-surface area on day 1. The EP regimen consisted of at most 6 cycles of etoposide 100 mg/m2 of body-surface area from day 1 to 3 and cisplatin 75mg/m2 of body-surface area on day 1. Cycle length for the two arms was 3 weeks. The dose adjustment was allowed in at most within ±5% per investigator discretion if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) of 0 to 2
* A life expectancy of at least 3 months
* Measurable lesions
* Adequate hematologic function

Exclusion Criteria:

* Infection
* Myocardial infarction within the preceding three months
* Symptomatic brain metastases or receiving radiotherapy less than 4 weeks
* Pregnancy or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, PhD, Principal Investigator — Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College; xingsheng Hu, Principal Investigator — Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China